CLINICAL TRIAL: NCT05238207
Title: A Phase Ia/Ib Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacodynamics of BBI-001 in Iron Deficient Volunteers and HH Patients
Brief Title: A Study to Evaluate BBI-001 in Hereditary Haemochromatosis (HH) Patients and Iron Deficient Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Only Part A (single dosing) was conducted due to business considerations
Sponsor: Bond Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBI001-101
Record Dates: First submitted 2022-01-24; First posted 2022-02-14 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Hereditary Hemochromatosis
MeSH Terms: conditions — Hemochromatosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BBI-001 (Experimental): BBI-001: Oral administration immediately prior to a meal enriched with stable iron isotope Fe57
  Interventions: Drug: BBI-001
- Placebo (Placebo Comparator): Placebo: Oral administration immediately prior to a meal enriched with stable iron isotope Fe58
  Interventions: Dietary Supplement: Original Fibre Metamucil

INTERVENTIONS:
Drug: BBI-001 — Part A: 1 dose BBI-001 administered in a crossover fashion Part B: 2 doses BBI-001 administered in a crossover fashion
  Arms: BBI-001
Dietary Supplement: Original Fibre Metamucil — Part A: 1 dose placebo administered in a crossover fashion Part B: 2 doses placebo administered in a crossover fashion
  Arms: Placebo

SUMMARY:
This is a first in human, double-blind, randomized, placebo-controlled, two-arm crossover study evaluating the safety, tolerability and PD of ascending dose levels of BBI-001 after:

* a single administration in iron deficient male and female participants, and male and female HH patients (Part A),
* two administrations per day in HH patients (Part B). BBI-001 administrations will be accompanied with consumption of a meal enriched with stable iron isotope Fe57, while corresponding placebo dose administrations will be with a meal enriched with stable iron isotope Fe58.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy iron deficient participants or patients with hereditary hemochromatosis

Exclusion Criteria:

* Serious or unstable medical or psychiatric conditions
* Significant medical history
* Current infections
* Receiving iron chelation therapy or treatment other than stable maintenance phlebotomy for the prior 6 months
* Organ damage from iron overload in the view of the PI would prevent successful completion of the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE) | up to 17 days
  Incidence, type, and severity of AEs, to include clinically significant laboratory changes
Clinical Laboratory Testing - Iron Panel | up to 17 days
  Changes from baseline in iron panel

SECONDARY OUTCOMES:
Evaluation of Iron Isotope Blood Levels | up to 17 days
  Fe57 and Fe58 blood concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Scribner, MD, Study Chair — Sponsor GmbH
Locations (1):
- Nucleus Networks, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No